CLINICAL TRIAL: NCT01533584
Title: Evaluation of Nocturnal Hypertension With 24-hour Ambulatory or Home Blood Pressure Measurement: Correlation With Target-Organ Damage
Brief Title: Evaluation of Nocturnal Hypertension and Correlation With Target-Organ Damage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George S. Stergiou, Associate Professor of Medicine and Hypertension, University of Athens
Other Study IDs: NOCTURNAL TOD
Record Dates: First submitted 2012-02-09; First posted 2012-02-15 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Nocturnal Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate nocturnal hypertension with 24-hour ambulatory blood pressure and home blood pressure (BP) measurements through a) comparison of mean BP and nocturnal dipping assessed with the two methods, b) correlation of those parameters with parameters of target-organ damage and c) comparison of the potential of the two methods to define non-dippers.

DETAILED DESCRIPTION:
It is well known that blood pressure (BP) exhibits diurnal variation. Nocturnal fall of BP normally exceeds 10%. Subjects with such fall of BP during sleep are classified as "dippers" and those with a nocturnal fall of BP less than 10% are classified as "non-dippers". Non-dippers are exposed to a greater cardiovascular risk. To date dipping status is defined with 24-hour ambulatory BP monitoring (ABPM). Many studies have shown that Home BP monitoring (HBPM) can be an alternative to daytime ambulatory BP monitoring and it exhibits similar correlation to markers of hypertension target-organ-damage (TOD). Nocturnal hypertension shows closer correlation with TOD, than daytime hypertension. In this study patients will be provided with a new-technology, reliable oscillometric device for HBPM, equipped with a modified algorithm, which allows scheduled automated BP measurements during sleep (Microlife WatchBP Home Nocturnal). Duplicate morning and evening BP measurements with one-minute interval will be performed by the patient sitting during seven working days. Afterwards a 24-hour ABPM will be performed, using Microlife WatchBP O3 oscillometric device, with a 20-minute interval between measurements. This order may be reversed according to the wish of the patient and devices' availability. Participants will visit site 3 times. Office blood pressure will be measured during two visits. Triplicate measurements with Microlife WatchBP Home Nocturnal will be performed at the sitting position.

TOD will be assessed with:

* cardiac triplex (LVMI)
* carotid triplex (ΙΜΤ)
* pulse wave velocity.
* Albumin/creatinine ratio measured in morning urine sample.

ELIGIBILITY:
Inclusion Criteria:

* Mean 24-hour Systolic BP (SBP) >130 mmHg and/or Mean 24-hour Diastolic BP (DBP) >80 mmHg.
* Patients physically and mentally capable of self-measuring BP at home.
* Written informed consent.

Exclusion Criteria:

* Sustained arrhythmia.
* Pregnancy.
* Symptomatic cardiovascular disease.
* Any other serious illness (cardiac, renal, or malignancy).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred for high Blood Pressure, untreated or, if treated for less than 2 weeks, 4 weeks after withdrwal of treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Hypertension Clinic, 3rd Dept. of Medicine, Evaggelismos Hospital., Athens
  - Hypertension Center, Third Department of Medicine, University of Athens, Greece, Athens